CLINICAL TRIAL: NCT01916187
Title: A Pilot Study of Imetelstat Given Intravenously on Day 1 and 8 of a 21 Day Schedule Alone and With Standard 13-Cis-Retinoic Acid in Children With Recurrent and/or Refractory Neuroblastoma
Brief Title: Imetelstat Given Intravenously Alone and With Standard 13-Cis-Retinoic Acid in Children With Neuroblastoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: drug company withdrew support following re-examination of benefit-risk assessment for the investigational use of imetelstat in this population
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: Geron Corporation (Industry)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I212
Record Dates: First submitted 2013-07-31; First posted 2013-08-05 (Estimated); Last update posted 2020-09-21 (Actual); Status verified 2020-04

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — imetelstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imetelstat (Experimental): 285 mg/m2/dose, IV, for 2 hours. Days 1 and 8 every three weeks.
  Interventions: Drug: Imetelstat

INTERVENTIONS:
Drug: Imetelstat

SUMMARY:
The purpose of this study is to determine the best dose of imetelstat when given alone for patients with neuroblastoma and also when given in combination with 13-cis-retinoic acid.

DETAILED DESCRIPTION:
This research is being done because imetelstat has been shown to slow the growth of tumours in animals and may also be doing so in adults, but we are not sure if it can also slow tumour growth in children and offer better results than standard treatment. Laboratory studies suggest imetelstat may increase the activity of 13-cis-retinoic acid, which is used to treat neuroblastoma, although this is not yet proven in patients.

ELIGIBILITY:
Inclusion Criteria:

* Histological verification of neuroblastoma at either original diagnosis or relapse.
* Patients must have recurrent or refractory neuroblastoma with either measurable or evaluable disease (defined by a positive nuclear scan such as bone scan or metaiodobenzylguanidine (MIBG) scan). If a lesion is isolated and /or previously irradiated and stable, a proven positive biopsy will be required to be eligible.
* Current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life.
* Must have recovered from the acute effects of prior chemotherapy, immunotherapy or radiotherapy prior to study entry as follows:

  * At least 3 weeks from completion of last active cancer therapy and recovered from toxic effects of that therapy to ≤ grade 1.
  * At least 6 weeks post hematopoietic stem cell rescue following myeloablative therapy.
  * At least 3 months must have elapsed if prior total body irradiation, craniospinal XRT or if ≥ 50% radiation of pelvis.
  * At least 6 weeks must have elapsed if other substantial bone marrow irradiation.
  * At least 6 weeks from prior MIBG therapy.
* Age >18 months and ≤18 years at the time of study entry.
* Performance Status:

Patients ≤10 years: Lansky ≥50 Patients >10 years: Karnofsky ≥60% - Laboratory Requirements: (must be done within 7 days prior to registration)

Adequate Bone Marrow Function, defined as:

* Absolute neutrophil count (ANC) ≥1.0 x 10^9/L
* Platelets ≥100 x 10^9/L (transfusion independent defined as not receiving platelet transfusions within 7 days prior to registration)
* Hemoglobin ≥80 g/L (may receive RBC transfusions) Patients with known bone marrow metastatic disease will be eligible for the study and may receive transfusions, provided ≤25% of bone marrow is involved, and provided they are not known to be refractory to red cell or platelet transfusions.

Patients will be eligible as long as blood count criteria are met. If patients then experience prolonged myelosuppression, bone marrow examination can be requested to determine if the low blood counts are due to malignant infiltration of the marrow or to therapy induced hypoplasia/aplasia.

Adequate Renal And Cardiac Function, defined as:

* Serum creatinine ≤1.5 x upper limit of normal for age or
* Measured GFR ≥70 mL/min/1.73 m2

Adequate Liver Function, defined as:

* AST and ALT ≤2.5 x upper limit normal for age
* Total bilirubin ≤1.5 x upper limit normal for age
* Serum albumin ≥ 20

Adequate Coagulation Function, defined as:

• PTT <1.2 x upper limit normal

* Patient or guardian consent must be obtained on all patients according to local Institutional and/or University Human Experimentation Committee requirements. Children > 8 years old whose parent or guardian has signed consent on their behalf may also sign assent if desired. It will be the responsibility of the local participating investigators to obtain the necessary local clearance, and to indicate in writing to the NCIC CTG Study Coordinator that such clearance has been obtained, before the trial can commence in that centre.
* Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits (for example: two hour's driving distance) placed on patients being considered for this trial.
* Protocol treatment is to begin within 5 working days of patient registration.

Exclusion Criteria:

* Patients with >25% bone marrow involvement will not be enrolled.
* Patients must be able to take oral medication and have no gastrointestinal abnormalities (e.g. bowel obstruction or previous gastric resection) which would lead to inadequate absorption of 13-cisretinoic acid.
* Known HIV, hepatitis B or hepatitis C infections.
* Imetelstat animal and in vitro studies suggest it is not genotoxic or teratogenic. However, 13-cis-retinoic acid is known to be teratogenic. Pregnancy tests must be obtained in girls who are post menarchal. Males or females of reproductive potential may not participate unless they have agreed to use two reliable contraceptive methods. Pregnant or breast-feeding females will not be entered on this study due to the potential fetal and teratogenic adverse effects.
* Concurrent Medications:

  * Patients receiving other investigational agents will not be enrolled.
  * Patient receiving other anti-cancer agents will not be enrolled.
  * Patients with CNS metastasis will need to submit to a baseline MRI obtained within 21 days prior to registration. Patients with evidence of current or prior CNS hemorrhage will be excluded. Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study will not be enrolled.

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07-30 (Actual); Primary Completion 2013-11-22 (Actual); Study Completion 2014-01-16 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Imetelstat in pediatric dose | 24 month
  Response and progression will be evaluated in this study using the revised international criteria (1.1) proposed by the RECIST (Response Evaluation Criteria in Solid Tumours) committee in patients with relapsed and/or refractory neuroblastoma, to confirm the feasibility of administering imetelstat given at the recommended pediatric dose as determined in the Children's Oncology Group Study ADVL1112 (a phase I study of imetelstat, a telomerase inhibitor, in children with recurrent or refractory solid tumours and lymphoma), alone and in combination with 13-cis-retinoic acid.

SECONDARY OUTCOMES:
Impact of imetelstat on hematopoietic stem cells and neuroblastoma tumour cells. | 24 months
  Bone marrow aspirates, biopsies and blood samples for CC assay: at baseline, end of cycles 1 and 2 then end of every other cycle will be assessed in patients with relapsed and/or refractory neuroblastoma to assess the impact of imetelstat on hematopoietic stem cells and neuroblastoma tumour initiating cells.
Changes in plasma C-circles | 24 months
  In patients with relapsed and/or refractory neuroblastoma to evaluate:
  * The correlation of tumour and plasma C-circles.
  * The role of plasma C-circles as a tumour biomarker for alternative lengthening of telomeres (ALT).
  * Changes in plasma C-circles induced by treatment with imetelstat.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Lewis, Study Chair — Alberta Children's Hospital, Southern Alberta Children's Cancer Program, AB Canada
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No